CLINICAL TRIAL: NCT03717506
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Comparison Study to Determine the Therapeutic Equivalence of GDC 268 and Clindamycin Phosphate Topical Lotion, 1% in Subjects With Acne Vulgaris
Brief Title: Bioequivalence Study of Clindamycin Phosphate Topical Lotion, 1% in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Balmoral Medical company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GDC-268-001
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Acne Vulgaris
Keywords: zits; pimples; blackheads
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test product (Experimental): GDC 268 Lotion applied topically as directed.
  Interventions: Drug: GDC 268 Lotion
- Reference Product (Active Comparator): Clindamycin Phosphate Lotion, 1% applied topically as directed.
  Interventions: Drug: Clindamycin Phosphate Lotion 1%
- Placebo (Placebo Comparator): GDC Vehicle lotion applied topically as directed.
  Interventions: Drug: GDC Vehicle Lotion

INTERVENTIONS:
Drug: GDC 268 Lotion — GDC 268 is a topical lotion
  Arms: Test product
Drug: Clindamycin Phosphate Lotion 1% — Clindamycin Phosphate Lotion is an FDA-approved drug product
  Arms: Reference Product
Drug: GDC Vehicle Lotion — GDC Vehicle Lotion contains 0.0% of active drug and is matched to the other two active test drugs
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the safety, tolerability, and therapeutic equivalence of GDC 268 to Clindamycin Phosphate Topical Lotion, 1% and to compare the efficacy of these two products to the GDC vehicle lotion (i.e., placebo) in the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female, ≥12 and ≤40 years of age with a clinical diagnosis of acne vulgaris.
* Must have ≥ 25 but ≤ 100 non-inflammatory lesions (open and closed comedones) AND ≥ 20 but ≤ 70 inflammatory lesions (papules and pustules) AND ≤ 2 nodulocystic lesions (nodules and cysts) on the face (e.g., forehead, nose, cheeks, chin, upper lip) at Baseline.
* Must be willing and able to refrain from use of all other topical products in the treatment area, all acne medications other than test article, and all antibiotics (other than test article) during the 12-week treatment period.
* Women must be surgically sterile, or use an effective method of birth control with a negative urine pregnancy test (UPT) at the Baseline Visit (Day 1).
* In good general health and free of any other clinically significant disease state or physical condition.
* Subject has provided written informed consent / assent.

Exclusion Criteria:

* Subject is pregnant, breastfeeding, or is planning to become pregnant or breastfeed during the study.
* Subject has more than 2 facial nodular lesions; any nodules present will be documented but not included in the inflammatory lesion count for analysis.
* Subject has excessive facial hair (e.g., beards, sideburns, moustaches), facial tattoos, or other facial attributes that would interfere with diagnosis or assessment of acne vulgaris in the opinion of the investigator.
* Subject is planning surgery during the study.
* Subject has a history of hypersensitivity or allergy to clindamycin or lincomycin and/or any of the ingredients in the test articles.

Other Eligibility Criteria not listed above will be reviewed for each prospective subject by the study staff.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1236 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Site 07, Fort Smith, Arkansas
  - Site 22, Rogers, Arkansas
  - Site 25, Fountain Valley, California
  - Site 33, Northridge, California
  - Site 30, San Diego, California
  - Site 44, Aventura, Florida
  - Site 36, Brandon, Florida
  - Site 45, DeLand, Florida
  - Site 41, Largo, Florida
  - Site 38, Miami, Florida
  - Site 35, Miami Lakes, Florida
  - Site 37, North Miami Beach, Florida
  - Site 26, St. Petersburg, Florida
  - Site 42, Tampa, Florida
  - Site 01, West Palm Beach, Florida
  - Site 10, Newnan, Georgia
  - Site 09, Boise, Idaho
  - Site 05, Rolling Meadows, Illinois
  - Site 02, Plainfield, Indiana
  - Site 27, Overland Park, Kansas
  - Site 28, Clarkston, Michigan
  - Site 24, Fridley, Minnesota
  - Site 49, Omaha, Nebraska
  - Site 06, High Point, North Carolina
  - Site 32, Raleigh, North Carolina
  - Site 19, Dublin, Ohio
  - Site 17, Gresham, Oregon
  - Site 34, Philadelphia, Pennsylvania
  - Site 20, Warwick, Rhode Island
  - Site 08, Anderson, South Carolina
  - Site 29, Chattanooga, Tennessee
  - Site 03, Murfreesboro, Tennessee
  - Site 04, Nashville, Tennessee
  - Site 43, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Product | Reference Product | Placebo
Started | 496 | 491 | 249
Completed | 447 | 441 | 222
Not Completed | 49 | 50 | 27

BASELINE CHARACTERISTICS:
Population: The baseline population includes the Safety and mITT populations, defined as all randomized subjects who applied at least one dose of the test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Placebo | Total
Number analyzed (Participants) | 496 | 491 | 249 | 1236
Age, Customized [Mean (Standard Deviation); unit: years] | 19.5 (6.4) | 19.3 (6.0) | 19.0 (5.1) | 19.3 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 287 | 287 | 151 | 725
  Male | 209 | 204 | 98 | 511
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 216 | 204 | 108 | 528
  Not Hispanic or Latino | 280 | 287 | 141 | 708
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Other category includes subjects that identified with more than one race.
  Participants
    Race: American Indian or Alaska Native | 2 | 2 | 0 | 4
    Race: Asian | 20 | 17 | 9 | 46
    Race: Black or African American | 119 | 114 | 54 | 287
    Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
    Race: White | 346 | 350 | 181 | 877
    Race: Other (multiple) | 8 | 8 | 4 | 20
Investigator's Global Assessment [Count of Participants; unit: Participants] — To be eligible for study participation, subjects required a clinical diagnosis of mild to severe facial acne vulgaris defined as Grade 2, 3, or 4 on the IGA at Baseline. The IGA (Investigator's Global Assessment) Scale is measured using a five-point scale from 0=Clear to 4=Severe.
  Participants
    2-Mild | 126 | 129 | 66 | 321
    3-Moderate | 332 | 319 | 172 | 823
    4-Severe | 38 | 43 | 11 | 92
Non-Inflammatory Lesions [Mean (Standard Deviation); unit: Lesions] | 44.9 (20.41) | 44.9 (19.31) | 45.5 (19.42) | 45.0 (19.77)
Inflammatory Lesions [Mean (Standard Deviation); unit: Lesions] | 28.3 (8.74) | 28.4 (9.55) | 27.7 (8.64) | 28.2 (9.05)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in the Number of Inflamed Lesions
Description: Percent Change from Baseline to Week 12 in inflammatory lesion counts (Papules/Pustules).
Time Frame: 12 weeks
Population: Analysis population is the per-protocol population defined as all subjects in the modified Intent-to-treat (mITT) population who met the following criteria: 1) Met all I/E criteria; 2) No evidence of material dosing noncompliance, 3) Completed the primary endpoint evaluation at Week 12 within the designated visit window (Day 85 ± 6 days), 4) Had no protocol violations that would affect the treatment evaluation, and 5) Did not use any prohibited medications.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Test Product | Reference Product | Placebo
Number analyzed (Participants) | 382 | 389 | 193
percent change | -39.4 (36.10) | -40.0 (36.83) | -35.1 (35.54)

2. Primary Outcome: Mean Percent Change in the Non-inflammatory Lesion Counts
Description: Percent Change (i.e., reduction) from Baseline to Week 12 in non-inflammatory (open and closed comedones) lesion counts.
Time Frame: 12 weeks
Population: Data based on the per-protocol population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Test Product | Reference Product | Placebo
Number analyzed (Participants) | 382 | 389 | 193
percent change | -52.7 (33.98) | -54.3 (34.44) | -43.0 (39.13)

3. Secondary Outcome: The Percentage of Subjects With a Clinical Response (IGA) of "Success" at Week 12
Description: Investigator's Global Assessment, IGA. Overall severity of acne was assessed using a five-point scale from 0=Clear to 4=Severe. Subjects must have had an IGA score of 2 (mild), 3 (moderate), or 4 (severe) at Baseline. Success is defined as an IGA score at week 12 that is at least 2 grades less than the baseline assessment.
Time Frame: 12 weeks
Population: Based on the per-protocol population.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | Reference Product | Placebo
Number analyzed (Participants) | 382 | 389 | 193
Participants | 78 | 64 | 18

4. Other Pre Specified Outcome: Incidence of Adverse Events
Description: Adverse Events (AEs) will be assessed by the investigator and the incidence (severity and causality) of any local and systemic AEs will be reported by number and percentage.
Time Frame: Day 1 through Day 85
Population: Based on the Safety population defined as all subjects randomized and applied at least one dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | Reference Product | Placebo
Number analyzed (Participants) | 496 | 491 | 249
Participants | 53 | 41 | 29

ADVERSE EVENTS:
Time Frame: 12 Weeks
Groups:
- Reference Product: Clindamycin Phosphate Lotion, 1% applied topically as directed.
  Clindamycin Phosphate Lotion 1%: Clindamycin Phosphate Lotion is an FDA-approved drug
Arm/Group | Test Product | Reference Product | Placebo
All-Cause Mortality (participants affected / at risk) | 0/496 | 0/491 | 0/249
Serious Adverse Events (participants affected / at risk) | 0/496 | 0/491 | 0/249
Other Adverse Events (participants affected / at risk) | 0/496 | 0/491 | 0/249

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 18 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 60 days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT03717506/Prot_SAP_000.pdf